CLINICAL TRIAL: NCT03588234
Title: Food Literacy and Type 1 Diabetes
Status: Completed | Type: Observational
Sponsor: McGill University (Other)
Collaborators: Diabetes Québec (Other)
Responsible Party: Principal Investigator, Anne-Sophie Brazeau, Assistant Professor, McGill University
Other Study IDs: 43-0618
Record Dates: First submitted 2018-07-04; First posted 2018-07-17 (Actual); Last update posted 2020-09-16 (Actual); Status verified 2020-09

CONDITIONS: Type1diabetes

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Type 1 diabetes: Individuals with type 1 diabetes (18-29 years old). They must complete a questionnaire. This group has approximately 26 extra questions to respond to compared to controls. The extra questions pertain to their diabetes history as well as their knowledge regarding diabetes.
- Matched controls without Type 1 diabetes: Individuals without type 1 diabetes (18-29 years old). They must complete the same questionnaire as the individuals with diabetes (without the diabetes-specific questions).

SUMMARY:
The objective of the current study is to assess the prevalence of poor food literacy in young adults with type 1 diabetes through a national on-line survey. More specifically, the research question to be investigated as part of this project is: What is the current level of food literacy among young adults with type 1 diabetes? It is hypothesized that at least 50% of young adults with type 1 diabetes have a poor level of food literacy.

DETAILED DESCRIPTION:
Food literacy, the ability to plan and manage, select, prepare, and eat healthy foods, is a contemporary concept that provides a mechanism to understand the relationship between food-related knowledge, skills (ie., culinary competencies) and health behaviours and its impact on decision-making regarding dietary intake. The Diabetes Canada 2018 Clinical Practice Guidelines have recognized the role that food skills, a component of food literacy, have in managing glycemic control in patients living with type 1 diabetes. The guidelines also point out that no studies to date have investigated this skill level in the diabetic population and that interventions aimed at improving these skills would be beneficial for patients. There is therefore a need to assess the current level of food literacy among young adults with type 1 diabetes in order for future studies to develop targeted interventions.

The project will be cross-sectional in design and data will be collected with an on-line questionnaire. This questionnaire will allow for the evaluation of the level of food literacy in young adults with and without type 1 diabetes. The online survey software that will be utilized is Survey Monkey.

The study will be publicized through posts on Facebook©, Twitter©, and other forms of social media as well as on websites of collaborating diabetes organizations (see appendix B for a list of organizations). Participants interested in the study will be invited to go on the survey webpage. The first information presented will be the electronic consent form. If they have questions while reading the consent form, they will have the possibility to email or call a research assistant. Once they have agreed, they will be re-directed to the first question. The questionnaire takes approximately 20-25 minutes to complete. Completion of the questionnaire will trigger a page requesting them to email the study coordinator in order to be entered into the lottery for a chance to win an Ipad mini.

The survey includes sociodemographic questions as well as medical and diet history. For participants with diabetes, this includes duration since their diabetes onset, types of treatments (insulin), application of carbohydrate counting and the "Type 1 Diabetes Nutrition Knowledge Survey". Items on actual food intake, such as fruits and vegetables, and self-efficacy regarding cooking are included. Food literacy will be evaluated using the "Short food literacy questionnaire (SQLF)", a short 12-item questionnaire that we adapted for Canada. A score for the SQLF will be calculated (maximum 52 points) and participants will be categorized under 4 different groups (Inadequate, Problematic, Sufficient, Excellent). Participants categorized in inadequate or problematic will be considered having low food literacy. Three questions regarding cooking ability were taken from the Canadian Community Health Survey (CCHS). Current sources of information regarding diet and nutrition, as well as questions to assess knowledge of chronic diseases linked to dietary intake, the frequency at which participants cook their own meals vs. eat out vs. consume prepackaged meals as well as specific dietary habits such as skipping breakfast will also be investigated. Lastly, perceived food environment will be assessed by asking questions regarding where participants shop for food and their satisfaction regarding the selection of food available to them.

ELIGIBILITY:
Inclusion Criteria:

* Type 1 diabetes

Ages: 18 Years to 29 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Young adults (18-29) with type 1 diabetes.
Sampling Method: Probability Sample
Enrollment: 427 (Actual)
Dates: Start 2018-06-28 (Actual); Primary Completion 2020-03-01 (Actual); Study Completion 2020-08-31 (Actual)

PRIMARY OUTCOMES:
Food literacy level | Baseline
  Short food literacy questionnaire (SFLQ) score. A score for the SQLF will be calculated (minimum score 7 points, maximum 52 points points) and participants will be categorized under 4 different groups (Inadequate, Problematic, Sufficient, Excellent). Participants categorized in inadequate or problematic will be considered having low food literacy.

SECONDARY OUTCOMES:
Fruit and vegetable consumption | Baseline
  On a daily basis, how many servings of fruits/vegetables do you eat on average?
Hypoglycaemia frequency | Baseline
  Overall, during a usual week, how many times does your blood sugar go low (lower than 4,0 mmol/L)?
Self-reported A1c | Baseline
  What was your last hemoglobin A1c result?
Fast food consumption | Baseline
  In the last week, how many times have you eaten at a fast food restaurant?

CONTACTS AND LOCATIONS:
Locations (1):
- McGill University, Montreal, Quebec, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Vidgen HA, Gallegos D. Defining food literacy and its components. Appetite. 2014 May;76:50-9. doi: 10.1016/j.appet.2014.01.010. Epub 2014 Jan 22. PMID 24462490
- [Background] Canadian Diabetes Association Clinical Practice Guidelines Expert Committee; Cheng AY. Canadian Diabetes Association 2013 clinical practice guidelines for the prevention and management of diabetes in Canada. Introduction. Can J Diabetes. 2013 Apr;37 Suppl 1:S1-3. doi: 10.1016/j.jcjd.2013.01.009. Epub 2013 Mar 26. No abstract available. PMID 24070926
- [Background] Fitzgerald JT, Funnell MM, Anderson RM, Nwankwo R, Stansfield RB, Piatt GA. Validation of the Revised Brief Diabetes Knowledge Test (DKT2). Diabetes Educ. 2016 Apr;42(2):178-87. doi: 10.1177/0145721715624968. Epub 2016 Jan 14. PMID 26769757
- [Background] Grea Krause C, Beer-Borst S, Sommerhalder K, Hayoz S, Abel T. A short food literacy questionnaire (SFLQ) for adults: Findings from a Swiss validation study. Appetite. 2018 Jan 1;120:275-280. doi: 10.1016/j.appet.2017.08.039. Epub 2017 Sep 11. PMID 28912107
- [Background] Statistics Canada, Canadian Community Health Survey (CCHS): Food skills - mechanical skills and food conceptualization. 2013: Ottawa.